CLINICAL TRIAL: NCT03201276
Title: Individual Differences in Glucosamine Sulfate Exposure Levels and Related Gene Polymorphism Research
Brief Title: Individual Differences in Glucosamine Sulfate Exposure Levels
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Qing Jiang, Vice Dean, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: glucosaminexzh
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Knee Osteoarthritis
Keywords: glucosamine sulfate; individual differences; gene polymorphism
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Drug group: patients taking glucosamine
  Interventions: Drug: Glucosamine Sulfate

INTERVENTIONS:
Drug: Glucosamine Sulfate — Patients taking glucosamine sulfate 1500mg every day for at least four days.

SUMMARY:
Glucosamine is an important part of the treatment strategy for osteoarthritis, but its effectiveness is still controversial. To explain the efficacy differences of glucosamine, in this study the investigators detect the concentration of glucosamine in the plasma and synovial fluid, some effect indexes such as inflammatory markers and gene polymorphism of glucosamine transporters. On the one hand, the investigators compare the plasma peak and gluten glucosamine concentration and the concentration in synovial fluid among participants to observe the individual differences of glucosamine exposure in vivo. On the other hand, the investigators investigate the correlation between drug concentrations, effect index and gene polymorphism. The hypothesis is that glucosamine exposure in vivo has individual differences and gene polymorphism can explain this differences.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing total knee arthroplasty for knee osteoarthritis;
2. 60-80 years.

Exclusion Criteria:

1. patients with severe liver or renal insufficiency;
2. patients allergic to glucosamine or any excipients in tablets;
3. patients who have been treated with glucosamine within three months;
4. patients who are unable to cooperate with the study;
5. continuous medication is less than 4 days;
6. patients with diarrhea, vomiting and other adverse reactions during medication.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee arthroplasty for knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-07-02 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Drug concentration in plasma | Fasting venous blood before the first administration
  Drug concentration is measured by HPLC-MS/MS
Drug concentration in plasma | 3 hours after the third administration
  Drug concentration is measured by HPLC-MS/MS
Drug concentration in plasma | 9 hours after the third administration
  Drug concentration is measured by HPLC-MS/MS
Drug concentration in plasma | Fasting venous blood before the fourth administration
  Drug concentration is measured by HPLC-MS/MS
Drug concentration in plasma | Venous blood during the operation of total knee arthroplasty
  Drug concentration is measured by HPLC-MS/MS
Drug concentration in synovial fluid | During the operation of total knee arthroplasty
  Drug concentration is measured by HPLC-MS/MS
Inflammatory markers in plasma | Fasting venous blood before the first administration
  Leptin
Inflammatory markers in plasma | 3 hours after the third administration
  Leptin
Inflammatory markers in plasma | 9 hours after the third administration
  Leptin
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  Leptin
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  Leptin
Inflammatory markers in plasma | Fasting venous blood before the first administration
  IL-1β
Inflammatory markers in plasma | 3 hours after the third administration
  IL-1β
Inflammatory markers in plasma | 9 hours after the third administration
  IL-1β
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  IL-1β
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  IL-1β
Inflammatory markers in plasma | Fasting venous blood before the first administration
  COX-2
Inflammatory markers in plasma | 3 hours after the third administration
  COX-2
Inflammatory markers in plasma | 9 hours after the third administration
  COX-2
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  COX-2
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  COX-2
Inflammatory markers in plasma | Fasting venous blood before the first administration
  IL-6
Inflammatory markers in plasma | 3 hours after the third administration
  IL-6
Inflammatory markers in plasma | 9 hours after the third administration
  IL-6
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  IL-6
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  IL-6
Inflammatory markers in plasma | Fasting venous blood before the first administration
  TNFα
Inflammatory markers in plasma | 3 hours after the third administration
  TNFα
Inflammatory markers in plasma | 9 hours after the third administration
  TNFα
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  TNFα
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  TNFα
Inflammatory markers in plasma | Fasting venous blood before the first administration
  MMP-3
Inflammatory markers in plasma | 3 hours after the third administration
  MMP-3
Inflammatory markers in plasma | 9 hours after the third administration
  MMP-3
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  MMP-3
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  MMP-3
Inflammatory markers in plasma | Fasting venous blood before the first administration
  ADAM-TS5
Inflammatory markers in plasma | 3 hours after the third administration
  ADAM-TS5
Inflammatory markers in plasma | 9 hours after the third administration
  ADAM-TS5
Inflammatory markers in plasma | Fasting venous blood before the fourth administration
  ADAM-TS5
Inflammatory markers in plasma | During the operation of total knee arthroplasty
  ADAM-TS5
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  Leptin
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  IL-1β
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  COX-2
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  IL-6
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  TNFα
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  MMP-3
Inflammatory markers in synovial fluid | During the operation of total knee arthroplasty
  ADAM-TS5
Gene polymorphism | Fasting venous blood before the first administration
  Gene polymorphisms of glucosamine transporters in vivo

REFERENCES:
- [Background] Chan PS, Caron JP, Orth MW. Effects of glucosamine and chondroitin sulfate on bovine cartilage explants under long-term culture conditions. Am J Vet Res. 2007 Jul;68(7):709-15. doi: 10.2460/ajvr.68.7.709. PMID 17605605
- [Background] Herrero-Beaumont G, Ivorra JA, Del Carmen Trabado M, Blanco FJ, Benito P, Martin-Mola E, Paulino J, Marenco JL, Porto A, Laffon A, Araujo D, Figueroa M, Branco J. Glucosamine sulfate in the treatment of knee osteoarthritis symptoms: a randomized, double-blind, placebo-controlled study using acetaminophen as a side comparator. Arthritis Rheum. 2007 Feb;56(2):555-67. doi: 10.1002/art.22371. PMID 17265490
- [Background] Setnikar I, Rovati LC. Absorption, distribution, metabolism and excretion of glucosamine sulfate. A review. Arzneimittelforschung. 2001 Sep;51(9):699-725. doi: 10.1055/s-0031-1300105. PMID 11642003